CLINICAL TRIAL: NCT02969824
Title: Post-acute Structured Exercise Following Sport Concussion: a Randomized Controlled Study
Brief Title: Post-acute Structured Exercise Following Sport Concussion
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated prematurely due to COVID pandemic in July 2020 in Toronto, Canada. Our institution did not allow for in-person research, making continuation of the study untenable.
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Michael Hutchison, Assistant Professor, Director, Concussion Program, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 33459
Record Dates: First submitted 2016-11-01; First posted 2016-11-21 (Estimated); Last update posted 2022-01-14 (Actual); Status verified 2021-12

CONDITIONS: Concussion, Brain
Keywords: Sport Injury; Concussion; Active Recovery
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care Group (No Intervention): Following a brief period of physical and cognitive rest (typically1-7 days, depending on symptom severity and timing of spontaneous symptom abatement), the physician advises participants to increase their activity levels gradually with minimal head movement (predominantly involving a stationary bike) and progressively increase levels of exertion while remaining under the threshold of symptom exacerbation. Subsequently, exercise progressed to include a progression of head movements, visual and cognitive burdens, sport-specific activities, and heavy resistance, in that order, all below the symptom exacerbation threshold.
- Supervised Exercise Group (Experimental): These individuals will begin to exercise at Day 3 post-injury. These participants will be asked to complete a total of eight exercise sessions over the course of 11 days, with one day of rest after two consecutive sessions. Two of the sessions (i.e., first and mid-point) will be an in-person exercise sessions at the lab with a member of the research team while the remaining six sessions will be home-based exercise sessions with remote communication by phone (i.e., call or text) with a member of the research team. Once individuals in this group achieve asymptomatic status, they will be directed through the existing return to play guidelines.
  Interventions: Behavioral: Supervised Aerobic Exercise

INTERVENTIONS:
Behavioral: Supervised Aerobic Exercise — The AE protocol will consist of eight sessions that proceed in a stepwise fashion in terms of duration and intensity over 11 days. Exercise will be performed on the Velotron Pro stationary cycle ergometer (RacerMate Inc., WA, USA), which will be digitally connected to a heart rate monitor and programmed to monitor the wattage of the bike based on the participant's heart rate. Exercise duration (15min-20min) and intensity (60%-75% max HR) will increase over the intervention period. For the remotely supervised sessions, exercise intensities and heart rate will be monitored via FitBit.
  Other Names: Exercise intervention
  Arms: Supervised Exercise Group

SUMMARY:
This study will investigate the effect of structured, standardized aerobic exercise (AE) compared to usual care on clinical recovery from sport-related concussion (SRC) within the post-acute phase of injury. Participants will be randomized into one of two groups: (1) Supervised Exercise Group: participants will complete a total of eight exercise sessions over the course of 11 days, starting at Day 3 post-injury (two sessions (first and mid-point) will be done in the lab, and the remained will be home-based sessions); (2) Usual Care Group: individuals will undergo a period of physical rest and standard care. For the purposes of this study, "rest" will be defined as the avoidance of any activities beyond those of daily living, including participation in sport and physical activity.

DETAILED DESCRIPTION:
A number of physical, cognitive, somatic, and emotional symptoms commonly occur following sports-related concussion. The most recent Concussion in Sport Consensus Statement recommends an initial period of rest (24-48 hours), followed by more activity - gradual and progressive - while staying below their cognitive and physical symptom-exacerbation thresholds. While structured exercise is advised post-injury, the appropriate intensity, frequency, and duration of activity remains unclear. Furthermore, there is also evidence that too much physical activity may be related to worse outcomes, which necessitates the investigation on the appropriate prescription of exercise following concussion.

Early work identified the potential benefit of exercise in those with persistent symptoms after concussion. However, it is important to recognize that exercise must be structured and tailored as it has been found that athletes engaging in high levels of activity post-injury were associated with greater symptom burden and poorer cognitive abilities. Collectively, these findings further support the potential benefit of personalized, prescribed exercise post-concussion.

Additional evidence in support of sub-acute and acute exercise interventions following neurological insult exists for other conditions of the central nervous system, such as low back pain, whiplash, and stroke. For example, research suggests that bed rest may actually delay recovery from acute low back pain, and recommendations to resume regular activities as soon as possible following injury result in faster recovery times, less chronic disability, and fewer recurrent problems. While rest and collar restraint were previously the standard mode of treatment for whiplash, recent evidence suggests that early mobilization and exercise compared to more traditional rest strategies. In terms of stroke, it has been shown that mobilization within 24 hours of this type of injury can expedite recovery while also inducing the risk of complications.

Therefore, the purpose of this study is to examine the effect of a structured, standardized, subacute AE intervention in adolescents after SRC, on time to recovery compared to usual care. This study will provide meaningful information regarding the utility of AE intervention after concussion. Findings from these works may inform future usual care procedures post-injury, potentially providing the first known treatment to improve recovery after concussion.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with SRC by a physician at the David L. MacIntosh Sport Medicine Clinic
* Minimum of 13 years of age and a maximum of 25 years of age
* Able to speak and understand English

Exclusion Criteria:

* Have had a previous concussion within two weeks of the presenting SRC
* Have any co-morbid injuries (i.e. musculoskeletal/soft-tissue injuries, vestibular disorders)
* Have a pre-existing heart condition
* Have any uncontrolled seizure disorders or a history of medical or neurological conditions that affects cognitive functioning

Ages: 13 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2017-02-16 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Clinical recovery - Days to Medical Clearance | Up to 1-year post-injury
  Number of days from the time of injury until a concussed athlete is cleared to return to play by a sport-medicine physician.

SECONDARY OUTCOMES:
Change in Symptoms | 28 Days: assessed at Days 7, 14, 21, 28, and 90 post-injury
  Concussion-related symptoms will be assessed using the Post-Concussion Symptom Scale (PCSS) of the Sport Concussion Assessment Tool-3 (SCAT3). The symptom score is comprised of a 22-item post-concussion symptom scale using a seven-point Likert scale rating. Total symptoms is the total number of symptoms with a non-zero score and symptom severity is obtained by summing the rated symptom score for each symptom.
Change in Heart Rate Variability (HRV) | 28 Days: assessed at Days 7, 14, 21, 28, and 90 post-injury
  Heart Rate Variability (HRV) will be assessed using the Polar heart rate V800 sports watch and corresponding chest strap heart monitor (Polar ®, QC, Canada). HRV will be assessed for 5 minutes in the supine position, followed by a 1-minute accommodation period, a final five-minute HRV assessment in the upright-seated position will be performed. HRV measurements to be analyzed HRV was assessed using both time domain and frequency domain measures, in accordance with recommendations of the Task Force of the European Society Cardiology and North American Society of Pacing and Electrophysiology.
Change in Blood Pressure Variability (BPV) | 28 days: assessed at Days 7, 14, 21, 28, and 90 post-injury
  Blood Pressure Variability (BPV) will be measured using the Finapres MIDI figure cuff device concurrently with HRV. Systolic BP and diastolic BP values will be acquired throughout the acquisition period.
Change in Peripheral Blood Biomarkers | 28 Days: assessed at Days 7, 14, 21, 28, and 90 post-injury
  Peripheral blood samples (approximately 20 mL) will be drawn from participants by a trained phlebotomist. High sensitivity multiplexed immunoassay will be employed to quantitate 30 inflammatory cytokines and chemokines, and 11 central nervous-injury specific biomarkers. Individual biomarker values will be excluded if they were above or below the manufacturers' recommended level of quantitation for each analyte, or displayed a coefficient of variance >25% between duplicates. Because multiple 96-well plates will analyzed, inter-plate variance will also be accounted for; therefore, plates will only be included in the statistical analysis if the inter-plate variance was <20%, calculated from internal control samples acquired on each plate. Raw values of biomarker analyte will be used in all analyses.
Change in Cognition | 28 Days: assessed at Days 7, 14, 21, 28, and 90 post-injury
  C3 Logix (iPad platform, Cleveland, OH, USA), will be employed to measure reaction time, information processing speed, visual acuity, and postural stability. This assessment will take approximately 10-15 minutes to complete. For each of subtest, the percent correct (accuracy) and reaction time (ms) will be analyzed.
Salivary MicroRNA and DNA Collection | 28 Days: assessed at Days 7, 14, 21, 28, and 90 post-injury
  A research team member will collect a very small amount of saliva (approximately 1mL) using a swab for MicroRNA analysis, and 2ml of liquid saliva for DNA analysis. This process normally takes approximately 3 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hutchison, PhD, Principal Investigator — University of Toronto
Locations (2):
- Canada (2):
  - David L. MacIntosh Sport Medicine Clinic, Toronto, Ontario
  - Goldring Centre for High Performance Sport, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be made available to other researchers. Study data will be retained for 10 years by the principal investigator, allowing adequate time for preparation and dissemination of research findings. All electronic files will be permanently deleted at the end of the retention period. De-identified data in the collective form may be made available to other researchers within our institution before this happens in order to generate more publications from this dataset. It may obtained by the principal investigator, who will maintain this data within a password-protected network.

REFERENCES:
- [Background] McCrory P, Meeuwisse W, Aubry M, Cantu B, Dvorak J, Echemendia RJ, Engebretsen L, Johnston K, Kutcher JS, Raftery M, Sills A; Kathryn Schneider, PT, PhD, Charles H. Tator, MD, PHD; Benson BW, Davis GA, Ellenbogen RG, Guskiewicz KM, Herring SA, Iverson G, Jordan BD, Kissick J, McCrea M, McIntosh AS, Maddocks DL, Makdissi M, Purcell L, Putukian M, Turner M, Schneider K, Tator CH. Consensus statement on concussion in sport--the 4th International Conference on Concussion in Sport held in Zurich, November 2012. Clin J Sport Med. 2013 Mar;23(2):89-117. doi: 10.1097/JSM.0b013e31828b67cf. No abstract available. PMID 23478784
- [Background] Silverberg ND, Iverson GL. Is rest after concussion "the best medicine?": recommendations for activity resumption following concussion in athletes, civilians, and military service members. J Head Trauma Rehabil. 2013 Jul-Aug;28(4):250-9. doi: 10.1097/HTR.0b013e31825ad658. PMID 22688215
- [Background] Thomas DG, Apps JN, Hoffmann RG, McCrea M, Hammeke T. Benefits of strict rest after acute concussion: a randomized controlled trial. Pediatrics. 2015 Feb;135(2):213-23. doi: 10.1542/peds.2014-0966. Epub 2015 Jan 5. PMID 25560444
- [Background] Dishman RK, Berthoud HR, Booth FW, Cotman CW, Edgerton VR, Fleshner MR, Gandevia SC, Gomez-Pinilla F, Greenwood BN, Hillman CH, Kramer AF, Levin BE, Moran TH, Russo-Neustadt AA, Salamone JD, Van Hoomissen JD, Wade CE, York DA, Zigmond MJ. Neurobiology of exercise. Obesity (Silver Spring). 2006 Mar;14(3):345-56. doi: 10.1038/oby.2006.46. PMID 16648603
- [Background] Marzolini S, Tang A, McIlroy W, Oh PI, Brooks D. Outcomes in people after stroke attending an adapted cardiac rehabilitation exercise program: does time from stroke make a difference? J Stroke Cerebrovasc Dis. 2014 Jul;23(6):1648-56. doi: 10.1016/j.jstrokecerebrovasdis.2014.01.008. Epub 2014 Apr 5. PMID 24709146
- [Background] Teasell RW, McClure JA, Walton D, Pretty J, Salter K, Meyer M, Sequeira K, Death B. A research synthesis of therapeutic interventions for whiplash-associated disorder (WAD): part 4 - noninvasive interventions for chronic WAD. Pain Res Manag. 2010 Sep-Oct;15(5):313-22. doi: 10.1155/2010/487279. PMID 21038010
- [Background] Hagen KB, Jamtvedt G, Hilde G, Winnem MF. The updated cochrane review of bed rest for low back pain and sciatica. Spine (Phila Pa 1976). 2005 Mar 1;30(5):542-6. doi: 10.1097/01.brs.0000154625.02586.95. PMID 15738787
- [Background] Baker JG, Freitas MS, Leddy JJ, Kozlowski KF, Willer BS. Return to full functioning after graded exercise assessment and progressive exercise treatment of postconcussion syndrome. Rehabil Res Pract. 2012;2012:705309. doi: 10.1155/2012/705309. Epub 2012 Jan 16. PMID 22292122
- [Background] Leddy JJ, Cox JL, Baker JG, Wack DS, Pendergast DR, Zivadinov R, Willer B. Exercise treatment for postconcussion syndrome: a pilot study of changes in functional magnetic resonance imaging activation, physiology, and symptoms. J Head Trauma Rehabil. 2013 Jul-Aug;28(4):241-9. doi: 10.1097/HTR.0b013e31826da964. PMID 23249769
- [Background] McCrory P, Meeuwisse W, Dvorak J, Aubry M, Bailes J, Broglio S, Cantu RC, Cassidy D, Echemendia RJ, Castellani RJ, Davis GA, Ellenbogen R, Emery C, Engebretsen L, Feddermann-Demont N, Giza CC, Guskiewicz KM, Herring S, Iverson GL, Johnston KM, Kissick J, Kutcher J, Leddy JJ, Maddocks D, Makdissi M, Manley GT, McCrea M, Meehan WP, Nagahiro S, Patricios J, Putukian M, Schneider KJ, Sills A, Tator CH, Turner M, Vos PE. Consensus statement on concussion in sport-the 5th international conference on concussion in sport held in Berlin, October 2016. Br J Sports Med. 2017 Jun;51(11):838-847. doi: 10.1136/bjsports-2017-097699. Epub 2017 Apr 26. No abstract available. PMID 28446457
- [Background] Carson JD, Lawrence DW, Kraft SA, Garel A, Snow CL, Chatterjee A, Libfeld P, MacKenzie HM, Thornton JS, Moineddin R, Fremont P. Premature return to play and return to learn after a sport-related concussion: physician's chart review. Can Fam Physician. 2014 Jun;60(6):e310, e312-5. PMID 24925965
- [Background] Williams RM, Puetz TW, Giza CC, Broglio SP. Concussion recovery time among high school and collegiate athletes: a systematic review and meta-analysis. Sports Med. 2015 Jun;45(6):893-903. doi: 10.1007/s40279-015-0325-8. PMID 25820456
- [Background] Waddell G, Feder G, Lewis M. Systematic reviews of bed rest and advice to stay active for acute low back pain. Br J Gen Pract. 1997 Oct;47(423):647-52. PMID 9474831
- [Background] Dahm KT, Brurberg KG, Jamtvedt G, Hagen KB. Advice to rest in bed versus advice to stay active for acute low-back pain and sciatica. Cochrane Database Syst Rev. 2010 Jun 16;2010(6):CD007612. doi: 10.1002/14651858.CD007612.pub2. PMID 20556780
- [Background] Schnabel M, Ferrari R, Vassiliou T, Kaluza G. Randomised, controlled outcome study of active mobilisation compared with collar therapy for whiplash injury. Emerg Med J. 2004 May;21(3):306-10. doi: 10.1136/emj.2003.010165. PMID 15107368
- [Background] Bernhardt J, Dewey H, Thrift A, Collier J, Donnan G. A very early rehabilitation trial for stroke (AVERT): phase II safety and feasibility. Stroke. 2008 Feb;39(2):390-6. doi: 10.1161/STROKEAHA.107.492363. Epub 2008 Jan 3. PMID 18174489
- [Derived] Hutchison MG, Di Battista AP, Lawrence DW, Pyndiura K, Corallo D, Richards D. Randomized controlled trial of early aerobic exercise following sport-related concussion: Progressive percentage of age-predicted maximal heart rate versus usual care. PLoS One. 2022 Dec 22;17(12):e0276336. doi: 10.1371/journal.pone.0276336. eCollection 2022. PMID 36548338